CLINICAL TRIAL: NCT04829864
Title: Phase 2 of STEP (Supporting the Transition to and Engagement in Parenthood): A Prenatal Intervention for Women Who Experienced Childhood Trauma
Brief Title: Supporting the Transition to and Engagement in Parenthood
Acronym: STEP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government); Social Sciences and Humanities Research Council of Canada (Other); Canada Research Chairs Endowment of the Federal Government of Canada (Other Government)
Responsible Party: Principal Investigator, Nicolas Berthelot, Professor, Université du Québec à Trois-Rivières
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STEP Phase 2
Record Dates: First submitted 2021-03-04; First posted 2021-04-02 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Trauma, Psychological; Prenatal Stress; Mental Health Issue; Maternal Distress
Keywords: Mentalization; Maternal bonding; Trauma; Well-being; Attachment; Pregnancy
MeSH Terms: conditions — Psychological Trauma; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEP (Experimental): Participants will participate, online or in-person, to the 8-9 sessions of the program addressing the psychological experience of pregnancy and supporting reflective capacities in relation to trauma and motherhood.
  Interventions: Behavioral: STEP
- Usual prenatal cares (No Intervention): Participants of the comparison group will receive usual prenatal cares (ex. prenatal classes)

INTERVENTIONS:
Behavioral: STEP — The program is offered by two facilitators to groups of three to seven women, in-person or online. The program is divided in three phases entitles "Becoming a mother"; "A look at my own history" and "Looking ahead". The first phase aims to explore and normalize the emotions experienced by the participants in the course of their pregnancy and to support the use of healthy emotion regulation strategies. The second phase aims to support mentalization of trauma, by discussing the nature of trauma and its impact; by validating participants' feelings as understandable responses to trauma; by supporting a reflection on positive and harsh experiences with significant others and the ways both types of experiences influenced participants' mental states; and identifying how participants coped with trauma. In the last phase, discussions focus on participants' needs and strengths, on available resources to support resilience and envision positive and challenging moments with the child.
  Arms: STEP

SUMMARY:
STEP (Supporting the Transition to and Engagement in Parenthood) is a manualized group intervention for pregnant women exposed to early life adversity designed to foster emotion regulation and reflective capacities in participants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages 18+ years
* Interested in reflecting about their experience of pregnancy and willing to attend weekly sessions in group setting.
* Must speak French as their first language

Exclusion Criteria:

* Severe psychiatric disorders (schizophrenia, bipolar disorder)
* Severe emotional dysregulation
* Current self-harm
* Not sure to keep the child
* High level of hostility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Change in psychological distress from baseline (2nd trimester of pregnancy) to the end of the third trimester of pregnancy (around 36 weeks) and from baseline to 6-months postpartum | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  Participants are invited to complete a self-report questionnaire (Kessler Distress Scale) assessing psychological distress. Change between baseline and end of pregnancy will be assessed, as well as between baseline and 6-month postpartum,
Perception of change in domains of functioning during pregnancy | Administered at one time-point, at the end of the third trimester of pregnancy. The participant will report on perceived changes during the last 9 months.
  We developed an instrument assessing one's perception of change (negative change to positive change) across multiple domains of functioning including the quality of the relationship with the partner; the quality of the relationship with significant others, self-esteem; emotion recognition, regulation and expression; social support and parental confidence. These domains will be assessed separately.
Level of satisfaction concerning the intervention | Satisfaction assessed after each session of the program and after its ending. Satisfaction is thus assessed between the second trimester of pregnancy and 36-weeks of pregnancy, for a total time frame up to 7-months.
  Participants are invited to complete a self-report questionnaire assessing their level of satisfaction after each session and at the end of the program, using a Likert scale. A semi-structured interview is also administered at the end of the program that will provide qualitative information regarding their appreciation of the program.
Prenatal reflective functioning | Administered at one time-point, at the end of the third trimester of pregnancy. The measure will assess current level of reflective functions.
  Participants will complete the Pregnancy Interview at the end of the third trimester of pregnancy. The interview will be subsequently coded for prenatal reflective functioning. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Parental reflective functioning | Administered at one time-point, at 6-moths postpartum. The measure will assess current level of reflective functions.
  Participants will complete the Parental Reflective Functioning Questionnaire at 6 months postpartum. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Change in trauma-specific reflective functioning | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  The Failure to mentalize trauma questionnaire (FMTQ) will be administered at baseline, at the end of the third trimester of pregnancy and at 6-months postpartum. Change between time-points will be assessed.
Change in trauma-specific reflective functioning | Administered at one time-point, at 6-moths postpartum. The measure will assess current level of reflective functions.
  Participants will participate to the Trauma Meaning Making Interview (TMMI) at 6-months postnatal. The interview will be subsequently coded for trauma-specific reflective functioning. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.

SECONDARY OUTCOMES:
Change in post-traumatic stress symptoms from baseline (2nd trimester of pregnancy) to the end of the third trimester of pregnancy (around 36 weeks) and from baseline to 6-months postpartum | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  Participants are invited to complete a self-report questionnaire of PTSD symptoms (Post-traumatic checklist for DSM-5). Change between baseline and the end of pregnancy will be assessed as well as between baseline and 6-months postpartum
Change in anger from baseline (2nd trimester of pregnancy) to the end of the third trimester of pregnancy (around 36 weeks) and from baseline to 6-months postpartum | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  Participants are invited to complete a self-report questionnaire of anger states (STAXI). Change between baseline and the end of pregnancy will be assessed as well as between baseline and 6-months postpartum
Change in perception of parental competence | Data will be collected at recruitment (2nd trimester of pregnancy) and at 36-weeks of pregnancy. The assessment time frame thus covers a period of 7 months.
  Participants are invited to complete a self-report questionnaire of maternal confidence (Maternal confidence questionnaire). Change between baseline and the end of pregnancy will be assessed.
Change in antenatal attachment | Data will be collected at recruitment (2nd trimester of pregnancy) and at 36-weeks of pregnancy. he assessment time frame thus covers a period of 7 months.
  Participants are invited to complete a self-report questionnaire of antenatal attachment (Maternal antenatal attachment scale). Change between baseline and the end of pregnancy will be assessed.
Self-compassion | Administered at one time-point, at the end of the third trimester of pregnancy. The measure will assess current level of self-compassion.
  Participants are invited to complete a self-report questionnaire of self-compassion at the end of the third trimester of pregnancy. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Connection to care | From the third trimester of pregnancy to 6 months postpartum. The assessment time frame thus covers a period of 7 months.
  Participants will be referred to community agencies for resources based on need during their participation to STEP. Their utilization of other resources will be assessed using self-reported questionnaires at the end of the third trimester of pregnancy and at 6 months postpartum
Change in emotion regulation strategies | Data will be collected at recruitment (2nd trimester of pregnancy) and at 36-weeks of pregnancy. he assessment time frame thus covers a period of 7 months.
  Participants are invited to complete a self-report questionnaire of emotion regulation strategies (CERQ). Change between baseline and the end of pregnancy, as well as between baseline and 6 months postpartum will be assessed.
Post-traumatic growth | Administered at one time-point, at the end of the third trimester of pregnancy. The measure will assess current level of post-traumatic growth.
  Participants are invited to complete a self-report questionnaire of post-traumatic growth at the end of the third trimester of pregnancy. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Parental stress | Administered at one time-point, at the 6-months postpartum assessment. The measure will assess current level of parental stress.
  Participants are invited to complete a self-report questionnaire of parental stress at 6-months postpartum. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Maternal bonding | Administered at one time-point, at the 6-months postpartum assessment. The measure will assess current level of maternal bonding.
  Participants are invited to complete a self-report questionnaire of maternal bonding at 6-months postpartum. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Maternal competence | Administered at one time-point, at the 6-months postpartum assessment. The measure will assess current level of perceived maternal competence..
  Participants are invited to complete a self-report questionnaire of maternal sense of competence at 6-months postpartum. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Depression | Data will be collected at 36-weeks of pregnancy and at 6-months postpartum. The assessment time frame thus covers a period of 7 months.
  Participants are invited to complete a self-report questionnaire of post-partum depression at the end of the third trimester of pregnancy and at 6-months postpartum. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention separately for each time point.
Maternal behaviors | Administered at one time-point, around 12-months postpartum. The measure will assess current maternal behaviors..
  Mother-infant interactions will be realized and videotaped for subsequent coding of maternal behaviors around 12-months postpartum. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention
Change in affective states from baseline (2nd trimester of pregnancy) to the end of the third trimester of pregnancy (around 36 weeks) and from baseline to 6-months postpartum | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  Participants are invited to complete a self-report questionnaire (Positive and Negative Affect Scale) assessing positive and negative affects. Change between baseline and end of pregnancy will be assessed as well as between baseline and 6-month postpartum,
Infant general development | Administered at one time-point, at 6-moths postpartum. The measure will assess current level of infant development.
  The ASQ-3 will be administered at 6-months postnatal to assess infant development.
Infant socio-emotional development | Administered at one time-point, at 6-moths postpartum. The measure will assess current level of infant development.
  The ASQ-SE will be administered at 6-months postnatal to assess infant socio-emotional development.
Infant temperament | Administered at one time-point, at 6-moths postpartum.The measure will assess current infant temperament
  The IBQ will be administered at 6-months postnatal to assess infant temperament

OTHER OUTCOMES:
Change in Inflammation | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  Inflammation will be assessed using blood samples at baseline, at the end of the third trimester of pregnancy and around 6 months postpartum. Change between baseline and the end of pregnancy, as well as between baseline and 6 months postpartum will be assessed.
Change in cortisol | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  Systemic cortisol will be assessed using blood samples at baseline, at the end of the third trimester of pregnancy and around 6 months postpartum. Change between baseline and the end of pregnancy, as well as between baseline and 6 months postpartum will be assessed.
Personality dysfunctions | Administered at one time-point, at the second trimester of pregnancy. The measure will assess current level of personality dysfunctions.
  Personality dysfunctions are assessed at baseline and will be considered as a moderator of the intervention effectiveness. Personality dysfunctions will be measured using the Self and Interpersonal Functioning Rating Scale, a 24-item self-report questionnaire designed to assess the four core elements of personality pathology (Identity, Self-direction, Empathy, and Intimacy) from the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Level of Personality Functioning for personality disorders
Change in intimate partner violence | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  Participants are invited to complete a self-report questionnaire of intimate partner violence. Change between baseline and 6 months postpartum will be assessed.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre intégré universitaire de santé et de services sociaux de la Capitale-Nationale, Québec, Quebec
  - Centre intégré de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.projetstep.ca
- See also: Related Info — http://www.stepproject.ca